CLINICAL TRIAL: NCT05107076
Title: Effect of PPCI on Diastolic Function & Levels of Galactin-3 in Patients With STEMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Bady Adly Hanna, Mariam Bady Adly Hanna, Assiut University
Other Study IDs: PPCI in STEMI patients
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Echocardiography; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STEMI patients who underwent PPCI: 2D Echocardiography with color Doppler assessment will be done within 24 h after PPCI
  Biochemical measurements:
  Peripheral blood samples were obtained within 48 hours after acute MI, and the serum will be frozen at -70°C until tested for Galactin-3 level.
  Follow up 2D Doppler echocardiography will be repeated at 40 days of the event.
  Interventions: Diagnostic Test: 2D Echocardiography with color Doppler assessment & Galactin-3 level in blood

INTERVENTIONS:
Diagnostic Test: 2D Echocardiography with color Doppler assessment & Galactin-3 level in blood — * Measurements will be
    1. Pulsed wave (PW) Doppler
    2. E (early diastolic)/A (late diastolic) - Using PW Doppler
    3. IVRT (isovolumic relaxation time)
    4. Deceleration time (DT) - from the peak of E wave to baseline.
    5. E/e'- PW tissue Doppler imaging (TDI)
    6. Left atrial volume and left atrial volume index (LAVI)
  * Peripheral blood samples will be obtained within 48 hours after acute MI, and the serum will be frozen at -70°C until tested for Galactin-3 level.

SUMMARY:
* 2D Echocardiography with color Doppler assessment: It will be done within 24 h after PPCI
* Peripheral blood samples were obtained within 48 hours after acute MI, and the serum will be frozen at -70°C until tested for Galactin-3 level.
* Follow up 2D Doppler echocardiography:

will be repeated at 40 days of the event.

DETAILED DESCRIPTION:
2D Echocardiography with color Doppler assessment:

It will be done within 24 h after PPCI. Measurements will be as following:

1. Pulsed wave (PW) Doppler will be performed in the apical 4chamber view within a 3 mm sample volume at the tip of the mitral leaflets to obtain mitral inflow velocities to assess LV filling.
2. E (early diastolic)/A (late diastolic) - Using PW Doppler, the peak E and A velocities were recorded, then the ratio of E/A will be calculated.
3. IVRT (isovolumic relaxation time) - derived by placing the cursor of Continuous wave (CW) Doppler in the LV outflow tract to simultaneously display the end of aortic ejection and the onset of mitral inflow.
4. Deceleration time (DT) - from the peak of E wave to baseline.
5. E/e'- PW tissue Doppler imaging (TDI) was performed in the apical views to acquire mitral annular velocities. The sample volume will be positioned at or 1 cm within the mitral leaflet's septal and lateral insertion sites.
6. Left atrial volume and left atrial volume index (LAVI) - The maximal left atrial (LA) volume measured from the apical four-chamber view using the modified Simpson method in end-systole before mitral valve opening. The LAVI obtained for all patients by dividing the LA volume by the body surface area.

Biochemical measurements:

Peripheral blood samples were obtained within 48 hours after acute MI, and the serum will be frozen at -70°C until tested for Galactin-3 level.

Follow up 2D Doppler echocardiography:

All previous echocardiographic measurements will be repeated at 40 days of the event.

ELIGIBILITY:
Inclusion Criteria:

* All patients of sample size admitted to the cardiology department of Assiut university hospital with:

  1. Acute typical chest pain
  2. Positive cardiac enzymes.
  3. ECG shows ST-segment elevation MI
  4. Documented occlusion of CA then treatment by PPCI

Exclusion Criteria:

* 1. Patients with well-known factors of left ventricular diastolic dysfunctions, including high blood pressure (over 140/90 mmHg), hypertrophic cardiomyopathy, left ventricular hypertrophy, bundle branch block, ventricular fibrillation, ventricular arrhythmia, severe valvular disease, complete heart block, and previous CABG.

  2. Patients with the end-stage renal disease usually have markedly increased galactin-3 levels 3. Prior use of thrombolytic agents 4. Refusal of PPCI due to social or religious concerns 5. ST elevation on ECG without obvious coronary artery diseases such as acute myocarditis, early repolarization, or Takotsubo cardiomyopathy 6. Atrial fibrillation at the time of echocardiography examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with age > 18 years who will present in the emergency department within 12 h (hrs) of the onset of ischemic chest pain & fulfill the diagnostic criteria of acute STEMI as defined by the universal definition of Myocardial Infarction (9) and are eligible for primary PCI will be included in this study.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Acute effect of PPCI in STEMI patients on diastolic function and Galactin-3 level | 48 hrs
  Determine the acute effect of PPCI in STEMI patients on the level of Galectin 3 and diastolic function within 48 hrs of the event.

SECONDARY OUTCOMES:
Correlation to patients' outcomes especially in those with initial high serum Galactin-3 | 40 days
  Correlating effect of PPCI on patients outcomes and impact on diastolic function, with consideration to those with initial high serum galectin levels at 40 days of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Helmy, Professor, Principal Investigator — Assiut University
Locations (1):
- Faculty of Medicine Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karaye KM, Sani MU. Factors associated with poor prognosis among patients admitted with heart failure in a Nigerian tertiary medical centre: a cross-sectional study. BMC Cardiovasc Disord. 2008 Jul 22;8:16. doi: 10.1186/1471-2261-8-16. PMID 18644161
- [Background] McManus DD, Chinali M, Saczynski JS, Gore JM, Yarzebski J, Spencer FA, Lessard D, Goldberg RJ. 30-year trends in heart failure in patients hospitalized with acute myocardial infarction. Am J Cardiol. 2011 Feb 1;107(3):353-9. doi: 10.1016/j.amjcard.2010.09.026. PMID 21256998